CLINICAL TRIAL: NCT06538376
Title: Clinical Utility of Portable Dynamic Chest X-Ray (DDR) in the ICU: Clinical Trial to Demonstrate the Feasibility of Deploying DDR Technology in the ICU - A Study to Prove Its Increased Diagnostic Value
Brief Title: Clinical Utility of Portable Dynamic Chest X Ray (DDR) in the ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Konica Minolta (Unknown)
Responsible Party: Principal Investigator, Gyorgy Frendl, M.D., Ph.D., Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023P001100
Record Dates: First submitted 2024-07-17; First posted 2024-08-05 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Edema; Pneumonia; Atelectasis; Pleural Effusion; Acute Rejection of Lung Transplant (Disorder); Airway Obstruction; Rib Fractures; Acute Copd Exacerbation; Asthma COPD; Pulmonary Embolism; Hemothorax; Pneumothorax; Mesothelioma; Diaphragmatic Paralysis
MeSH Terms: conditions — Pulmonary Edema; Pneumonia; Pulmonary Atelectasis; Pleural Effusion; Airway Obstruction; Rib Fractures; Pulmonary Embolism; Hemothorax; Pneumothorax; Mesothelioma; Respiratory Paralysis

STUDY DESIGN:
Intervention Model Description: All participants enrolled in the study will receive the same intervention- there are not separate control and intervention groups. The intervention is a new portably dynamic digital radiography (DDR) scan and will be compared to the patients clinically indicated gold standard diagnostic test (i.e. portable chest x-ray, VQ scan, CT, CT-angio, etc.).
Masking Description: The outcomes assessors (radiologists) will evaluate deidentified DDR scans and deidentified traditional x-rays for all study patients in a blinded fashion, and will not be able to compare readings of or diagnoses from each scan for individual patients until after the analysis is complete.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Portable Dynamic Digital Radiography (DDR) + Clinical Gold Standard Imaging (Experimental): Dynamic digital radiography (DDR) is a new version of chest radiography from Konica Minolta (KM) that provides more advanced measures of lung motion, ventilation, and perfusion compared to traditional chest radiography. DDR scans are dynamic images that have a rate of 15 frames per second (for 7-20 seconds), acting as a mini-fluorography machine with radiation that is only slightly greater than a traditional chest x-ray.
  Every patient will receive both a DDR scan and a gold standard scan. Each patient's DDR images will be compared to the golden standard that is completed as part of the patient's routine standard of care. For instance, for many ICU patients this includes traditional chest x-rays, ultrasounds or VQ scans.
  Interventions: Diagnostic Test: Portable Dynamic Digital Radiography (DDR)

INTERVENTIONS:
Diagnostic Test: Portable Dynamic Digital Radiography (DDR) — (DDR imaging has already been described in the arm/group description). Each patient in the study will receive at least one set of DDR images, which consists of one 7-second scan in which the patient breaths normally, and a second 7-second scan in which the patient holds their breath (or for ventilated patients, an inspiratory pause is placed by the care team).
  If the patient's conditions warrant it, up to two sets of follow-up scans may be acquired. For instance, in a patient with diaphragmatic dysfunction, imaging may be completed pre- and post- diaphragmatic plication.

SUMMARY:
Dynamic digital radiography (DDR) is a new advanced version of chest radiography that captures dynamic images at a rate of 15 frames per second. It is coupled with an analytical software that allows it to provide more advanced measures of lung motion, ventilation, and perfusion compared to traditional chest radiography. While implementation of DDR fixed machines are beginning elsewhere in the US, this trial involves the first applications of an FDA-approved portable DDR machine, for use at the bedside in the ICU.

The goal of this clinical trial is to determine the feasibility and safety of portable DDR technology in the ICU, as well as to evaluate the improved clinical diagnostic value of the portable DDR system over current standards of care.

Participants will receive one to three sets of DDR images, which will then be compared to their clinical gold standard exams (such as chest x-rays, CTs, or VQ scans) to assess and improve the precision and accuracy of measurements such as diaphragmatic motion, lung movement, and perfusion.

DETAILED DESCRIPTION:
Chest radiography was introduced to medical practice over a century ago, shortly after the discovery of X-rays by Roentgen. Since then, it has been a key component of the health, screening, clinical evaluation, and the assessments of therapy for billions of people. To this day, chest radiography remains the most frequently ordered imaging test. In this 700-bed tertiary care hospital, over 100,000 chest radiographs are obtained annually. The technique of chest radiography has remained largely unchanged and is seen as a mostly qualitative rather than quantitative tool. Chest dynamic X-ray (DDR) is a new advanced version of chest radiography that provides important quantitative parameters such as lung motion, ventilation, and perfusion. With a dynamic scan of 20-30 seconds, sequential images of both lungs are obtained with high temporal resolution during breathing (7.5-30 frames per second), without increasing radiation dose. DDR utilizes a dynamic digital radiography (DDR) technique with a flat-panel detector (2-6) and generates images with a field-of-view (FOV) that can cover both lungs. DDR utilizes detectors with higher sensitivity than those typically used in conventional radiography, enabling multiple dynamic time frames to be obtained despite keeping the dose mostly unchanged. Compared to conventional radiography, computer analysis and image processing of the DDR sequential time frames provide additional valuable metrics that capture motion and other key functions of the lungs, while high-quality chest radiographs can also be generated from the recombined frames. Chest DDR can be performed in essentially any patient position, including standing or sitting, to capture lung physiology in a manner representative of daily life. Furthermore, DDR is inexpensive, requires minimal space, and enables high throughput, which can help reduce medical costs. While area-detector CT can provide a higher temporal resolution, its FOV cannot entirely cover both lungs and its radiation dose can be prohibitively high. Chest DDR offers a unique opportunity to provide dynamic imaging parameters for lung motion and function in a safe, practical, and cost-effective manner.

Recently, the portable DDR technology has become available. This portable DDR scanner enables applications for non-mobile patients, like ICU patients. It allows the semi-quantitative or quantitative evaluation of pulmonary perfusion, ventilation, and diaphragmatic motion. ICU patients may have limited access to CT or MRI scanners due to the severity of their condition and/or to difficulties associated with support their devices (ECMO, LVAD, etc.), hence, why the portable DDR technology could have an especially meaningful impact on their care. The current Radiology team consists of Drs. Nishino, Wada, Valtchinov and Madore. The PI's group from Radiology will work in close collaboration with Dr. Frendl's research team in the BWH ICUs, as well as their biostatistician as multidisciplinary team of experts. They will also continue cooperation with Mr. Tsunomori and Mr. Yoneyama. These team members already have an established track record of successful collaboration with the PI.

The investigators will use the observational study design where two diagnostic imaging modalities will be compared for their ability to best diagnose lung pathologies (i.e., diaphragmatic motion and lung aeration/ventilation, pulmonary perfusion, and lung water content). These imaging modalities are: (i) the current portable AP chest x-ray (CXR)-based diagnostic technique and (ii) the recently developed portable dynamic chest XR (DDR) technique.

The DDR technology has yet to be proven to provide specific benefits for the care of the patients through the improved diagnosis of their pulmonary issues. Its ability to provide clinically meaningful additional information on aspects of lung pathologies (diaphragmatic motion and lung aeration/ventilation, pulmonary perfusion, and lung water content), that cannot be clearly discerned from the current portable CXR-based diagnostic technique, need to be documented; hence, the aims.

This study design will compare the ability to diagnose those lung pathologies (atelectasis, pulmonary embolus, and pulmonary edema) as determined by either the DDR technology or the traditional qualitative portable routine AP CXR (the current standards of diagnosis) through images obtained via the two techniques at the same time points for each patient. The DDR imaging and analysis will provide both qualitative and semi-quantitative data for each patient at all time points.

For this study, the patient's routine portable CXR will serve as the control image when applicable, and DDR images will serve as study images for each timepoint. For certain clinical conditions, the applicable gold standards will be used as controls, i.e. CT angiogram for pulmonary embolus, V-Q scans for lung ventilation and perfusion, and fluorographic swallowing studies for speech and swallow evaluation.

Data derived from these studies will be expected to provide novel and clinically crucial (quantitative or semi-quantitative) information on the degree of diaphragmatic excursion when the patient is spontaneously ventilating vs. when ventilator support is provided. This would be crucial for decision making regarding the patient's readiness for extubation, or, inversely, when poor excursion of the diaphragms is detected for non-ventilated patients, it would support the decision for early implementation of ventilator support. Data on lung aeration would also factor into this decision-making process.

Currently, quantitative or semi-quantitative data regarding these physiologic functions of the lungs are not available. Hence, why the investigators will focus on validating these novel metrics against clinical scenarios and outcomes. The investigators anticipate that this novel technology will better guide clinical decision making like the need for (or inversely, the safe removal of) ongoing ventilator support for our patients.

Furthermore, the perfusion (blood flow assessment) component of the image analysis would provide invaluable (currently unavailable) diagnostic options for those patients for whom CT angiogram is not available to rule out/confirm pulmonary embolism (PE). CT angiogram is not available for patients who suffer from hemodynamic instability, or when it is clinically contraindicated, like patients with impending renal failure. The added value of the DDR technology for the diagnosis of larger PEs will be assessed in the later stages of this study.

ELIGIBILITY:
Inclusion Criteria: Participants must meet all the following inclusion criteria to participate in this study:

* Adults (at least 18 years of age) including both intubated/ventilated and non-intubated patients
* Likely to have pathology related to either, abnormal diaphragmatic excursion and lung aeration, pulmonary perfusion, increased lung water content or all the above, as well as for cricopharyngeal dysfunction/swallowing difficulties at risk for aspiration.
* The subject or a legally authorized representative has provided written informed consent.

Exclusion Criteria: Candidates meeting any of the exclusion criteria at baseline will be excluded from study participation. These criteria are:

* Special populations, including women with known pregnancy, prisoners, or institutionalized individuals
* Patients where additional radiation is clinically contraindicated
* Care team does not provide assent for approaching patient/surrogate
* For women of child-bearing potential, defined as premenopausal women, a pregnancy test will be administered to determine pregnancy status and confirm eligibility for the study. A pregnancy test will NOT be administered to women who are post-menopausal or have documentation of surgical sterilization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
I. Extended clinical trial to study the degree of precision of the Portable DDR technology in assessing the cardiopulmonary functions of diaphragm and lung motion. | Up to 2 months
  Hypothesis: The Portable DDR technology can improve the visualization of parameters associated with lung physiology for ICU patients (diaphragmatic motion, lung motion) compared to current standards of care for imaging.
  Aim I-1: Determine the diagnostic precision of Portable DDR technology vs. routine standard of care imaging for specific lung pathologies (for example in pre- and post-transplant patients) that affect the mentioned cardiopulmonary functions.
  The DDR's precision will be measured by using the most relevant diagnostic procedure, the gold standard, for the condition will be used as reference to assess both qualitative and semiquantitative or quantitative information yielded by both types of imaging.
  The golden standard images for each of these parameters are:
  1. Diaphragmatic/Lung motion: Ultrasound imaging.
II. Extended clinical trial to study the degree of precision of the Portable DDR technology in assessing the cardiopulmonary functions of pulmonary blood flow. | Up to 2 months
  Hypothesis: The Portable DDR technology can improve the visualization of parameters associated with lung physiology for ICU patients (pulmonary blood flow) compared to current standards of care for imaging.
  Aim II-1: Determine the diagnostic precision of Portable DDR technology vs. routine standard of care imaging for specific lung pathologies (for example in pre- and post-transplant patients) that affect the mentioned cardiopulmonary function.
  The DDR's precision will be measured by using the most relevant diagnostic procedure, the gold standard, for the condition will be used as reference to assess both qualitative and semiquantitative or quantitative information yielded by both types of imaging.
  The golden standard image for this parameter is:
  1. Pulmonary blood flow: VQ scan or pulmonary angiograms
  The comparisons in precision for both diaphragm/lung motion and pulmonary blood flow will be aggregated to determine overall precision of the DDR technology

CONTACTS AND LOCATIONS:
Overall Officials: Gyorgy Frendl, MD PhD, Principal Investigator — Brigham and Women's Hospital; Hiroto Hatabu, MD PhD, Principal Investigator — Brigham and Women's Hospital; Bruno Madore, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Hata A, Yamada Y, Tanaka R, Nishino M, Hida T, Hino T, Ueyama M, Yanagawa M, Kamitani T, Kurosaki A, Sanada S, Jinzaki M, Ishigami K, Tomiyama N, Honda H, Kudoh S, Hatabu H. Dynamic Chest X-Ray Using a Flat-Panel Detector System: Technique and Applications. Korean J Radiol. 2021 Apr;22(4):634-651. doi: 10.3348/kjr.2020.1136. Epub 2020 Nov 30. PMID 33289365
- [Background] Fyles F, FitzMaurice TS, Robinson RE, Bedi R, Burhan H, Walshaw MJ. Dynamic chest radiography: a state-of-the-art review. Insights Imaging. 2023 Jun 19;14(1):107. doi: 10.1186/s13244-023-01451-4. PMID 37332064
- [Background] Ce M, Oliva G, Rabaiotti FL, Macri L, Zollo S, Aquila A, Cellina M. Portable Dynamic Chest Radiography: Literature Review and Potential Bedside Applications. Med Sci (Basel). 2024 Feb 7;12(1):10. doi: 10.3390/medsci12010010. PMID 38390860
- [Background] Yamada Y, Ueyama M, Abe T, Araki T, Abe T, Nishino M, Jinzaki M, Hatabu H, Kudoh S. Time-Resolved Quantitative Analysis of the Diaphragms During Tidal Breathing in a Standing Position Using Dynamic Chest Radiography with a Flat Panel Detector System ("Dynamic X-Ray Phrenicography"): Initial Experience in 172 Volunteers. Acad Radiol. 2017 Apr;24(4):393-400. doi: 10.1016/j.acra.2016.11.014. Epub 2016 Dec 15. PMID 27989446
- [Background] Hida T, Yamada Y, Ueyama M, Araki T, Nishino M, Kurosaki A, Jinzaki M, Honda H, Hatabu H, Kudoh S. Time-resolved quantitative evaluation of diaphragmatic motion during forced breathing in a health screening cohort in a standing position: Dynamic chest phrenicography. Eur J Radiol. 2019 Apr;113:59-65. doi: 10.1016/j.ejrad.2019.01.034. Epub 2019 Jan 31. PMID 30927960
- [Background] Yamada Y, Ueyama M, Abe T, Araki T, Abe T, Nishino M, Jinzaki M, Hatabu H, Kudoh S. Difference in diaphragmatic motion during tidal breathing in a standing position between COPD patients and normal subjects: Time-resolved quantitative evaluation using dynamic chest radiography with flat panel detector system ("dynamic X-ray phrenicography"). Eur J Radiol. 2017 Feb;87:76-82. doi: 10.1016/j.ejrad.2016.12.014. Epub 2016 Dec 16. PMID 28065378
- [Background] Hida T, Yamada Y, Ueyama M, Araki T, Nishino M, Kurosaki A, Jinzaki M, Honda H, Hatabu H, Kudoh S. Decreased and slower diaphragmatic motion during forced breathing in severe COPD patients: Time-resolved quantitative analysis using dynamic chest radiography with a flat panel detector system. Eur J Radiol. 2019 Mar;112:28-36. doi: 10.1016/j.ejrad.2018.12.023. Epub 2019 Jan 4. PMID 30777216